CLINICAL TRIAL: NCT04504851
Title: Rosuvastatin Evaluation as a Tuberculosis Treatment Adjunct
Acronym: ROSETTA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROSETTA
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Pulmonary Tuberculosis
Keywords: Statin; Rosuvastatin
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Rosuvastatin Calcium; Rifampin; Isoniazid; Pyrazinamide; Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Standard of Care) (Active Comparator): Standard combination treatment for pulmonary TB of 8 weeks rifampicin, isoniazid, pyrazinamide, ethambutol, then 16 weeks rifampicin, isoniazid
  Interventions: Drug: Rifampicin; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Ethambutol
- Arm B (Standard of Care plus Rosuvastatin) (Experimental): Standard combination treatment for pulmonary TB of 8 weeks rifampicin, isoniazid, pyrazinamide, ethambutol PLUS rosuvastatin, then 16 weeks rifampicin, isoniazid
  Interventions: Drug: Rosuvastatin 10mg; Drug: Rifampicin; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Ethambutol

INTERVENTIONS:
Drug: Rosuvastatin 10mg — 10mg of Rosuvastatin in the Intensive Phase of Therapy (8 weeks)
  Other Names: Crestor
  Arms: Arm B (Standard of Care plus Rosuvastatin)
Drug: Rifampicin — Rifampicin 10mg/kg
Drug: Isoniazid — Isoniazid 5mg/kg
Drug: Pyrazinamide — Pyrazinamide 25mg/kg
Drug: Ethambutol — Ethambutol 15mg/kg

SUMMARY:
This trial aims to determine whether the addition of rosuvastatin to standard TB therapy in pulmonary tuberculosis results in accelerated of sputum culture conversion. The trial will also investigate potential new biomarkers of sterilising activity and immune-modulatory activity.

DETAILED DESCRIPTION:
Rosuvastatin is an HMG Co-A reductase inhibitor which may be of value as possible adjunctive agents to standard TB therapy. Cell culture assays and animal models demonstrate that statins are bactericidal against Mtb with effects that are additive to that of anti-tuberculous therapy.

This is a Phase IIb randomised, controlled, open-label, early bactericidal activity trial. We will recruit patients between the ages of 18 and 75 with newly-diagnosed smear or Xpert positive pulmonary TB, who have had no more than 7 days of TB therapy.

Patients will be randomised to take either standard TB therapy or standard TB therapy plus rosuvastatin for the first 8 weeks of their therapy. After the first 8 weeks, patients will continue standard combination TB therapy and remain in trial follow-up until week 24. The trial will collect sputum for culture on a weekly basis for the first 8 weeks of the trial, and less frequently leading up to week 24.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 - 75 years of age
2. Abnormalities on CXR compatible with pulmonary TB
3. At least one sputum specimen, produced at or prior to screening during the current illness episode, that is:

   (i) positive for acid-fast bacilli on smear microscopy (with at least 1+ on the IUATLD/WHO scale) and/or (ii) positive on testing by Xpert MTB/RIF or Xpert Ultra (with semi-quantitative cycle threshold (CT) result of 'medium' or 'high')
4. Able to produce at least 5ml of sputum per day at the time of screening
5. Current or planned treatment with a regimen containing rifampicin, isoniazid and pyrazinamide (with or without ethambutol) only
6. Resident at a fixed address within feasible travelling distance to the site and likely to remain a local resident for the duration of trial follow-up
7. Willing to have directly observed therapy (DOT)
8. Willing to comply with the study visits and procedures

Exclusion Criteria:

1. More than 7 days of standard TB treatment by the time of the baseline visit
2. Known rifampicin resistance or isoniazid resistance at the time of randomization (results by conventional DST or molecular tests are not required to be available prior to randomization)
3. Previous treatment for active TB disease, unless rifampicin susceptibility has been demonstrated on a molecular test performed during this episode.
4. Extrapulmonary TB that, in the opinion of the treating clinician, is likely to require concurrent use of steroids, or require surgical management.
5. Known hypersensitivity to rosuvastatin
6. History of myopathy or family history of hereditary muscular disorders
7. Acute liver failure or decompensated chronic liver disease
8. Current alcohol abuse
9. Known hypothyroidism
10. Any of the following laboratory parameters at screening:

    1. ALT >3 times upper limit of normal (ULN)
    2. Estimated glomerular filtration rate (eGFR) < 60ml/min/1.73m2 (calculated using the CKD-EPI equation) (81)
    3. Creatine Kinase >5 times ULN
    4. Potassium <2.5 mmol/L
11. Active malignancy on chemotherapy or radiotherapy
12. Current use of immunosuppressive medication (≤ 5mg/ day of prednisolone or equivalent is acceptable).
13. HIV infection (unless patient has been stable on continuous antiretroviral therapy for at least 6 months, with CD4 count >/= 250 cells/mm3 and viral load </= 200 copies/ml, on a test performed at screening or during the last 12 months prior to screening, in which case they may be enrolled)
14. Use of any statin drug at screening or during the 3 months prior to screening
15. History of Atherosclerotic Cardiovascular Disease (ASCVD; defined as myocardial infarction, stable or unstable angina, coronary artery disease or coronary or other arterial revascularization, stroke, transient ischemic attack, or peripheral artery disease including aortic aneurysm, all of atherosclerotic origin)
16. Known Familial Hypercholesterolaemia
17. Other reasons, in the opinion of the investigator (and taking into consideration current local and international guidelines for primary prevention of cardiovascular disease), why the patient should commence statin treatment during the 6-month period following randomization
18. Current use of drugs contraindicated for use with rosuvastatin or standard TB drugs including fusidic acid, gemfibrozil, feno-fibrate, nicotinic acid (>1 gram/day), cyclosporine, directly acting antivirals for chronic Hepatitis C, protease inhibitors for HIV and praziquantel.
19. Women who are pregnant or breastfeeding
20. Women of childbearing potential unwilling or unable to use appropriate effective contraception for the first 12 weeks of the trial.
21. Any serious condition suggestive of myopathy or predisposing to the development of renal failure secondary to rhabdomyolysis (such as extensive surgery, significant trauma, uncontrolled seizures)
22. Any other severe underlying condition that would, in the opinion of the investigator, compromise the patient's safety or outcome in the trial.
23. Participation in other clinical intervention trial or research protocol (participation in other studies that do not involve an intervention may be allowed, but this must be discussed and approved by the Chief Investigator).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2020-08-12 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Time to culture conversion in Liquid Media | within 8 weeks after randomisation
  Time to culture conversion is defined is time from randomisation to the first of two consecutive negative sputum cultures

SECONDARY OUTCOMES:
Time to culture conversion in Solid media | within 8 weeks after randomisation
  Time to culture conversion is defined is time from randomisation to the first of two consecutive negative sputum cultures
Time to culture conversion in Liquid media | within 12 weeks after randomisation
  Time to culture conversion is defined is time from randomisation to the first of two consecutive negative sputum cultures
Sputum culture negative in Liquid media | at 8 weeks from randomisation
Sputum culture negative in Solid media | at 8 weeks from randomisation
Change in time to positivity (TTP) | from baseline to week 8
Change in proportion of lung affected on CXR | from baseline to week 8
Change in the aggregate cavity size on CXR | from baseline to week 8
Change in score on St George's Respiratory Questionnaire (SGRQ) | from baseline to week 8
Change in FEV1/FVC | from baseline to week 8
One or more Grade 3 or Grade 4 adverse events | by week 24
One of more Serious Adverse Events (SAEs) | by week 24

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Paton, Principal Investigator — National University Hospital, Singapore
Locations (6):
- Philippines (3):
  - Tropical Disease Foundation, Makati City
  - De La Salle Health Sciences Institute, Manila
  - Lung Center Philippines, Quezon City
- National University Hospital, Singapore, Singapore, Singapore
- Joint Clinical Research Centre, Kampala, Uganda
- Vietnam Military Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cross GB, Sari IP, Burkill SM, Yap CW, Nguyen H, Quyet D, Dalay VB, Gutierrez E, Balanag VM, Castillo RJ, Chang CC, Kelleher AD, O'Doherty J, Paton NI. PET-CT outcomes from a randomised controlled trial of rosuvastatin as an adjunct to standard tuberculosis treatment. Nat Commun. 2024 Dec 2;15(1):10475. doi: 10.1038/s41467-024-54419-3. PMID 39622823
- [Derived] Cross GB, Sari IP, Kityo C, Lu Q, Pokharkar Y, Moorakonda RB, Thi HN, Do Q, Dalay VB, Gutierrez E, Balanag VM, Castillo RJ, Mugerwa H, Fanusi F, Kwan P, Chew KL, Paton NI; ROSETTA trial team. Rosuvastatin adjunctive therapy for rifampicin-susceptible pulmonary tuberculosis: a phase 2b, randomised, open-label, multicentre trial. Lancet Infect Dis. 2023 Jul;23(7):847-855. doi: 10.1016/S1473-3099(23)00067-1. Epub 2023 Mar 23. PMID 36966799